CLINICAL TRIAL: NCT02861001
Title: Prospective, Randomized Study in Ventilated Critically Ill Patients Receiving Percutaneous Tracheotomy. A Comparison of Periinterventional Visualization of Conventional Bronchoscopy and an Endotracheal Tube Mounted Camera (VivaSight-SL™)
Brief Title: VivaSight-SL™ Versus Bronchoscopy for Percutaneous Tracheotomy
Acronym: VivaPDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VivaPDT
Record Dates: First submitted 2016-06-13; First posted 2016-08-10 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Insufficiency
Keywords: tracheotomy; bronchoscopy; critical care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bronchoscopic guidance (Active Comparator): optical guidance of percutaneous tracheotomy is done by conventional bronchoscopy
  Interventions: Device: conventional bronchoscopy
- tube mounted camera guidance (Experimental): optical guidance of percutaneous tracheotomy is done by the VivaSight-SL tube
  Interventions: Device: VivaSight-SL tube

INTERVENTIONS:
Device: conventional bronchoscopy — optical guidance of percutaneous tracheotomy is done by conventional bronchoscopy
  Arms: bronchoscopic guidance
Device: VivaSight-SL tube — optical guidance of percutaneous tracheotomy is done by the VivaSight-SL tube
  Arms: tube mounted camera guidance

SUMMARY:
Optical guidance for percutaneous tracheotomy in intensive care is usually performed by bronchoscopy. Recently, an endotracheal tube with a camera mounted at its tip (VivaSight-SL) has been introduced that allows for endotracheal visualization.

For feasibility evaluation, ten patients in intensive care receive percutaneous tracheotomy with optical guidance by the VivaSight-SL tube. If this part is completed with satisfactory results, patients are randomized to receive optical guidance by bronchoscopy or by VivaSight-SL tube. The primary end point is the visualization through the tube camera of endotracheal landmark structures for tracheotomy and visualization of the needle insertion (according to score, see detailed description).

DETAILED DESCRIPTION:
Background

Long-term ventilated critically ill patients often receive a tracheotomy to facilitate weaning from the ventilator and for prevention of secondary complications by the endotracheal tube [1]. Besides surgical tracheotomy in which a muco-cutaneous fistula is prepared between trachea and outer skin, percutaneous tracheotomy (PDT) has been introduced, in which a cannula is being inserted into the trachea. After introduction of a guidewire, the trachea is then dilated [2]. This intervention should be led by optical guidance, i. e. to verify the correct point of tracheal cannulation between the 2nd and 3rd tracheal cartilage and to minimize the risk for accidental injury to the membranous part of the trachea [3]. Usually, optical guidance is performed by bronchoscopy [4]. During bronchoscopy in ventilated patients, a drop in minute ventilation or an increase of carbon dioxide partial pressure with a consecutive respiratory acidosis may occur. Recently, an endotracheal tube with an integrated camera at its tip has been introduced that permits a continuous visualization of the trachea on a monitor connected to the camera (VivaSightTM-SL, ETView Ltd., Misgav, Israel) [5]. This tube has been CE and FDA certified (http://www.etview.com/products/ vivasight-sl).

In this study, it is being evaluated whether the optical guidance during PDT can be performed by the VivaSightTM-SL tube. Without the need for bronchoscopy during intervention, patients' ventilation during the procedure may be optimized with a lesser increase of the arterial and the end-expiratory carbon dioxide partial pressures. Furthermore, the procedure itself would be simpler without the need for a bronchoscopy.

In the investigators' institution, the VivaSightTM-SL tube has already been used in two patients together with bronchoscopic guidance for percutaneous tracheotomy. According to the investigators' experience, it seems to be possible to perform the procedure without a bronchoscopy. Therefore, the feasibility of PDT with guidance by the VivaSightTM-SL tube alone without bronchoscopy is tested. After a positive result in the first part of this study, non-inferiority of the VivaSightTM-SL tube in comparison to bronchoscopy is tested.

Methods

Design of Study / No. of Patients:

part 1: observational study, 10 consecutive patients part 2: randomized, prospective study, 46 patients

With a sample size of 46 (randomized 1:1 in 2 groups of 23 each) a difference of 35% on a visualization score [6] may be seen with an α-error of 0,05 and a β-error of 1-0,8.

Procedures:

* screening of for study inclusion according to inclusion and exclusion criteria
* changing of the endotracheal tube to the VivaSightTM-SL tube
* percutaneous tracheotomy with Ciaglia Blue Rhino technique [2, 7, 8]
* arterial blood gas sampling (BGA): baseline value from patients' records, prior to skin incision, immediately after insertion of tracheal tube

study inclusion:

All patients being treated in the Dept. of Intensive Care Medicine receiving percutaneous tracheotomy due to long term ventilation are screened according to inclusion and exclusion criteria.

Details of study-procedures:

Intubation:

The Intubation with the VivaSightTM-SL endotracheal tube does not differ from an intubation with a conventional tube that is done with respect to the standard operating procedure (SOP) of the Dept. for Intensive Care Medicine. During the intubation, vital parameters are monitored with respect to the underlying disease and patients' therapy is continuously adjusted. According to the SOP, two physicians are present of which at least one is a fellow or an attending physician with experience in intensive care medicine.

bronchoscopy:

The bronchoscopy for percutaneous tracheotomy is done according to the SOP of the Dept. for Intensive Care Medicine. Furthermore, during this study the bronchoscopy is done by a physician with an experience of more that 200 bronchoscopies.

percutaneous tracheotomy:

The tracheotomy is performed according to the Ciaglia Blue Rhino method [2, 7, 8] (Ciaglia Blue Rhino® G2, Cook Medical, Bloomington, IN, USA). After skin incision and an optional blunt dissection of the subcutaneous tissue, the trachea is cannulated between the 2nd and 3rd tracheal cartilage. Visualization is provided by either the VivaSightTM-SL tube or by conventional bronchoscopy. Should visualization be insufficient (one item of score ≥ 3, see below), a bronchoscope is available as a back-up. The tracheotomy is performed by an experienced fellow or attending physician.

rating of visualization of tracheal structures and ventilation during percutaneous dilatational tracheostomy (mod. after [6]):

Rating (each item 1 to 4 points)

A) Identification of: thyroid cartilage, cricoid cartilage, 1st-3rd tracheal cartilage

1 Reliable identification; 2 Only cricoid cartilage and tracheal cartilages; 3 Only tracheal cartilages; 4 No vision on tracheal structures

B) Visualization of tracheal circumference 1 Complete; 2 circumference 1/3 to 2/3 of circumference; 3 Only small parts of trachea; 4 No vision on tracheal structures

C) Monitoring puncture: midline + level below 1st or 2nd tracheal cartilage

1 Reliable identification; 2 Midline sure Level uncertain, but below the 1st tracheal cartilage; 3 Level of puncture uncertain; 4 No vision on tracheal structures

D) Monitoring dilatation Anterior wall and Pars membranacea (P.m.) visible; 1 Reliable identification; 2 P.m. only; 3 Only small parts of trachea visible, no control of P.m.; 4 No vision on tracheal structures

E) Quality of Ventilation Before puncture and worst ventilation during PDT, respectively

1 Minute ventilation (MV) as before starting tracheotomy; 2 MV < 2 L/min or oxygen saturation (SO2) 80-90% (>2minutes); 3 MV < 0,5l /min or SO2 70 - 79% (> 2 minutes); 4 MV = 0 or SO2 < 70% (> 2 minutes)

Consent: all patients or their legal surrogate give written informed consent.

Data protection: Data are anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving percutaneous tracheotomy in the Dept. of Intensive Care Medicine.
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Age < 18 years
* No consent
* Direct laryngoscopy according to Cormack-Lehane ≥ 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
visualization through the tube camera of endotracheal landmark structures for tracheotomy and visualization of the needle insertion (according to score) | during tracheotomy

SECONDARY OUTCOMES:
minute ventilation according to score generated from 4 point Likert scale at 2 time points | two time points: 1. during identification of landmark structures before puncture of trachea, 2. during puncture, dilatation and tracheotomy
pulse oxymetric oxygen saturation according to score generated from 4 point Likert scale at 2 time points | two time points: 1. during identification of landmark structures before puncture of trachea, 2. during puncture, dilatation and tracheotomy
change in pH-values | three time points: baseline value (up to 1h before tracheotomy), 0 min before skin incision, and 0 min before insertion of tracheal cannula
change in paCO2 values | three time points: baseline value (up to 1h before tracheotomy), 0 min before skin incision, and 0 min before insertion of tracheal cannula
  change in arterial partial pressure of carbon dioxide (mmHg)
change in etCO2 values | three time points: baseline value (up to 1h before tracheotomy), 0 min before skin incision, and 0 min before insertion of tracheal cannula
  change in endtidal carbon dioxide (mmHg)
change in paO2 values | three time points: baseline value (up to 1h before tracheotomy), 0 min before skin incision, and 0 min before insertion of tracheal cannula
  change in arterial partial pressure of oxygen (mmHg)
changes in peak airway pressure of ventilator | three time points: baseline value (before sterile drapes are applied), 0 min before skin incision, and 0 min before insertion of tracheal cannula
  if volume controlled mode is used
duration of the intervention | during tracheotomy
adverse events | up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, PhD, Principal Investigator — Head of Dept. of Intensive Care Medicine
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dreher M, Kluge S. [Airway devices in the intensive care unit]. Pneumologie. 2014 Jun;68(6):371-7. doi: 10.1055/s-0034-1365318. Epub 2014 Mar 25. German. PMID 24668495
- [Background] Ciaglia P, Firsching R, Syniec C. Elective percutaneous dilatational tracheostomy. A new simple bedside procedure; preliminary report. Chest. 1985 Jun;87(6):715-9. doi: 10.1378/chest.87.6.715. PMID 3996056
- [Background] Braune S, Kluge S. [Percutaneous dilatational tracheostomy]. Dtsch Med Wochenschr. 2011 Jun;136(23):1265-9. doi: 10.1055/s-0031-1280549. Epub 2011 May 31. No abstract available. German. PMID 21630175
- [Background] Vargas M, Sutherasan Y, Antonelli M, Brunetti I, Corcione A, Laffey JG, Putensen C, Servillo G, Pelosi P. Tracheostomy procedures in the intensive care unit: an international survey. Crit Care. 2015 Aug 13;19(1):291. doi: 10.1186/s13054-015-1013-7. PMID 26271742
- [Background] Huitink JM, Koopman EM, Bouwman RA, Craenen A, Verwoert M, Krage R, Visser IE, Erwteman M, van Groeningen D, Tijink R, Schauer A. Tracheal intubation with a camera embedded in the tube tip (Vivasight() ). Anaesthesia. 2013 Jan;68(1):74-8. doi: 10.1111/anae.12065. Epub 2012 Nov 5. PMID 23121322
- [Background] Linstedt U, Zenz M, Krull K, Hager D, Prengel AW. Laryngeal mask airway or endotracheal tube for percutaneous dilatational tracheostomy: a comparison of visibility of intratracheal structures. Anesth Analg. 2010 Apr 1;110(4):1076-82. doi: 10.1213/ANE.0b013e3181d27fb4. PMID 20357150
- [Background] Baumann HJ, Kemei C, Kluge S. [Tracheostomy in the intensive care unit]. Pneumologie. 2010 Dec;64(12):769-76. doi: 10.1055/s-0030-1255743. Epub 2010 Sep 20. German. PMID 20857374
- [Background] Byhahn C, Wilke HJ, Halbig S, Lischke V, Westphal K. Percutaneous tracheostomy: ciaglia blue rhino versus the basic ciaglia technique of percutaneous dilational tracheostomy. Anesth Analg. 2000 Oct;91(4):882-6. doi: 10.1097/00000539-200010000-00021. PMID 11004042
- [Derived] Grensemann J, Eichler L, Kahler S, Jarczak D, Simon M, Pinnschmidt HO, Kluge S. Bronchoscopy versus an endotracheal tube mounted camera for the peri-interventional visualization of percutaneous dilatational tracheostomy - a prospective, randomized trial (VivaPDT). Crit Care. 2017 Dec 29;21(1):330. doi: 10.1186/s13054-017-1901-0. PMID 29284503